CLINICAL TRIAL: NCT05875831
Title: Comparison Of Coughing and Active Cycle of Breathing Technique to Improve Pulmonary Functions in Post-Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/543
Record Dates: First submitted 2023-03-18; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Post Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coughing (Other)
  Interventions: Diagnostic Test: Coughing
- Active Cycle of Breathing (Experimental)
  Interventions: Behavioral: Active Cycle of Breathing

INTERVENTIONS:
Behavioral: Active Cycle of Breathing — Active Cycle of Breathing Technique to Improve Pulmonary Functions in Post-Surgical Patients
  Arms: Active Cycle of Breathing
Diagnostic Test: Coughing — Coughing to Improve Pulmonary Functions in Post-Surgical Patients
  Arms: Coughing

SUMMARY:
To find out the Comparison Of Coughing and Active Cycle of Breathing Technique to Improve Pulmonary Functions in Post-Surgical Patients

ELIGIBILITY:
Inclusion Criteria:

* Both male and female between the age of 18-50 years who reported post-surgical complications related to pulmonary will be selected in this study

Exclusion Criteria:

* If patient is unresponsive, psychologically disturbed and does not want to participate, teenagers will be excluded from this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Spirometry-related questions | 6 Months
surgical Related Questioner | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No